CLINICAL TRIAL: NCT02525263
Title: A Phase II, Open-label Safety and Efficacy Study of an Autologous Neo-Kidney Augment (NKA) in Patients With Type 2 Diabetes and Chronic Kidney Disease
Brief Title: Autologous Neo-Kidney Augment (NKA) in Patients With Type 2 Diabetes and Chronic Kidney Disease (CKD)
Acronym: RMCL-CL001
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The single patient enrolled began hemodialysis treatments.
Sponsor: Prokidney (Industry)
Collaborators: CTI Clinical Trial and Consulting Services (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RMCL-CL001
Record Dates: First submitted 2015-07-30; First posted 2015-08-17 (Estimated); Results first posted 2021-04-23 (Actual); Last update posted 2021-04-23 (Actual); Status verified 2021-03

CONDITIONS: Chronic Kidney Disease; Type 2 Diabetes
Keywords: Neo-Kidney Augment; Type 2 Diabetes; Chronic Kidney Disease; Cell Therapy
MeSH Terms: conditions — Renal Insufficiency, Chronic; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Neo-Kidney Augment (Experimental): NKA is made from expanded autologous selected renal cells (SRC) obtained from the patient's kidney biopsy. To manufacture NKA, kidney biopsy tissue from each enrolled patient will be sent to RegenMedTX, LLC, where renal cells will be expanded and SRC selected. SRC will be formulated in a gelatin based hydrogel at a concentration of 100 x 106 cells/mL, packaged in a 10 mL syringe, and shipped to the clinical site for use.
  Interventions: Biological: Neo-Kidney Augment

INTERVENTIONS:
Biological: Neo-Kidney Augment — NKA is made from expanded autologous selected renal cells (SRC) obtained from the patient's kidney biopsy. To manufacture NKA, kidney biopsy tissue from each enrolled patient will be sent to RegenMedTX, LLC, where renal cells will be expanded and SRC selected. SRC will be formulated in a gelatin based hydrogel at a concentration of 100 x 106 cells/mL, packaged in a 10 mL syringe, and shipped to the clinical site for use.

SUMMARY:
A Phase II, Open-Label Safety and Efficacy Study of an Autologous Neo-Kidney Augment (NKA) in Patients With Type 2 Diabetes and Chronic Kidney Disease (RMTX-CL001). NKA is made from expanded autologous selected renal cells (SRC) obtained from the patient's kidney biopsy. All enrolled subjects will be treated with up to two injections of NKA at least 6 months apart.

DETAILED DESCRIPTION:
A Phase II, Open-Label Safety and Efficacy Study of an Autologous Neo-Kidney Augment (NKA) in Patients With Type 2 Diabetes and Chronic Kidney Disease (RMTX-CL001). This is a Multi-center, prospective, open-label, single-group study. NKA is made from expanded autologous selected renal cells (SRC) obtained from the patient's kidney biopsy. To manufacture NKA, kidney biopsy tissue from each enrolled patient will be sent to RegenMedTX, LLC, where renal cells will be expanded and SRC selected. SRC will be formulated in a gelatin based hydrogel at a concentration of 100 x 106 cells/mL, packaged in a 10 mL syringe, and shipped to the clinical site for use. All enrolled subjects will be treated with up to two injections of NKA at least 6 months apart. Up to 30 subjects undergoing NKA injection will be enrolled into the study. Patients who have received a single injection of NKA under previous research protocols may enroll in this clinical trial to receive a single additional implantation. Patients who have never received an NKA injection may enroll in this clinical trial for up to a total of two (2) NKA injections, temporally spaced at least 6 months apart. All biopsies are to be taken from a single kidney, and all NKA injections are to be given into the kidney that was biopsied.

Patients who complete screening procedures satisfying all I/E criteria will be enrolled into the study immediately prior to the injection. Patients who do not meet all criteria before injection will be considered screen failures. Once a patient has been injected, the patient will have completed treatment and every effort should be made to ensure the patient completes all follow-up visits. Injection dates for the first 3 patients receiving their second NKA injection will be staggered by a minimum of 3 week intervals to allow for assessment of acute adverse events and other safety parameters by a Data Safety Monitoring Board (DSMB). At the completion of the follow-up visits, patients will continue in a long-term observational follow-up period. Patients will be followed for a total of 36 months following the last NKA injection under this protocol, whether the first or second injection.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females, age 30 - 70 years.
2. Patients with type 2 diabetes mellitus (T2DM).
3. Patients with diabetic nephropathy as the underlying cause of their renal disease.
4. If not previously implanted with NKA, CKD defined as a GFR of 20 - 50 mL/min/1.73m2 inclusive. Ifs previously treated with a single NKA implantation, eGFR 15 to 60 mL/min may also enroll.
5. Microalbuminuria (urinary albumin-creatinine ratio (UACR) ≥ 30 mg/g or urine albumin excretion ≥ 30 mg/day on 24 hour urine collection) not explained by an alternative diagnosis.
6. Systolic blood pressure between 105 and 140 mmHg (inclusive) and diastolic blood pressure ≤90 mmHg.
7. Treatment with angiotensin inhibitor (ACEI) or angiotensin blocker (ARB) initiated at least 8 weeks prior to enrollment. Treatment must be stable for the 6 weeks prior to implant. Patients intolerant of ACEI or ARBs may be included if stable BP is within acceptable limits.
8. Minimum of 2 measurements of eGFR or serum creatinine (sCr) at least 3 months apart and within 12 months before Screening, to define the rate of progression of CKD.
9. Willing and able to refrain from use of non-steroidal drugs (NSAIDs) (including aspirin), clopidogrel, fish oil, dipyridamole, prasugrel, or platelet inhibitors for 7 days before and after both biopsy and implant.
10. Willing and able to cooperate with all aspects of the study.
11. Willing and able to give signed informed consent.

Exclusion Criteria:

1. Type 1 diabetes mellitus (DM).
2. History of renal transplant.
3. HbA1c > 10% at Screening.
4. Hemoglobin levels < 9 g/dL prior to implant.
5. Known allergy to kanamycin or structurally similar aminoglycoside antibiotics.
6. Abnormal coagulation status as measured by partial thromboplastin time (APTT), international normalized ratio (INR), and/or platelet count at Screening.
7. Not a good candidate for the implantation procedure (based on the assessment of the investigator or operator) including patients who are morbidly obese, have BMI > 45, have excessive fat surrounding the kidney, or who are otherwise at risk for serious complications.
8. Clinically significant infection requiring parenteral antibiotics within 6 weeks of implantation.
9. Patients with small kidneys (average size < 9 cm) or only one kidney, as assessed by MRI or renal US within 1 year of screening.
10. Patients with acute kidney injury or a rapid decline in renal function within 3 months prior to implantation.
11. Patients with renal tumors, polycystic kidney disease, renal cysts or other anatomic abnormalities that would interfere with implantation procedure (e.g., cysts in the pathway of the injection for implantation), hydronephrosis, skin infection over proposed implantation sites, or evidence of a urinary tract infection.
12. Female subjects who are pregnant, lactating (breast feeding) or planning a pregnancy during the course of the study, or who are of child bearing potential and not using a highly effective method of birth control (including sexual abstinence). Subjects must be willing to continue birth control methods throughout the course of the study.
13. History of cancer within the past 3 years (excluding non-melanoma skin cancer and carcinoma in situ of the cervix).
14. Life expectancy of less than 2 years.
15. Any contraindication or known anaphylactic or severe systemic reaction to either human blood products or materials of animal (bovine, porcine) origin or anesthetic agents.
16. Positive for Human Immunodeficiency Virus (HIV), Hepatitis B Virus (HBV), or Hepatitis C Virus (HCV) assessed at the Screening Visit.
17. Subjects requiring treatment for tuberculosis (TB) in the past 3 years.
18. Immunocompromised subjects or patients receiving systemic immunosuppressive agents (including patients treated for chronic glomerulonephritis) within 3 months of implantation.
19. Subjects with uncontrolled diabetes (defined as metabolically unstable by the PI), or with incapacitating cardiac and/or pulmonary disorders.
20. History of active alcohol and/or drug abuse that in the investigator's assessment would impair the subject's ability to comply with the protocol.
21. Patients with elevated transaminases (ALT or AST > 3.0 x ULN) at Screening.
22. Patients with bleeding disorders that would, in the opinion of the Investigator, interfere with the performance of study procedures; patients taking coumarins (e.g. Warfarin) or other anticoagulants (e.g. enoxaparin or direct thrombin inhibitors).
23. Any circumstance in which the investigator deems participation in the study is not in the subject's best interest.
24. Use of any investigational product within 3 months of the implantation without receiving prior written consent of the Medical Monitor.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2016-07; Primary Completion 2017-05 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ashley Johns, MSHS, Study Director — Prokidney
Locations (1):
- University of North Carolina- Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The one US patient who had previously received an NKA injection under a previous protocol for the previous sponsor was allowed to enroll in this trial.
Pre-assignment Details: The only enrolled patient was assigned to the only treatment arm. There was no significant event prior to assignment.
Groups:
- NKA Augment Second Dose: This was an open-label, single treatment art trial. A previously treated patient was enrolled in this trial to be administered a second dose of NKA via the percutaneous route.
Period: Overall Study
Arm/Group | NKA Augment Second Dose
Started | 1 (The single patient in this trial was enrolled on 18 July 2016.)
Completed | 1 (The trial was completed when the patient reached the specified endpoint of starting hemodialysis.)
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The single US patient who had previously received an NKA injection was enrolled in this clinical trial.
Groups:
- NKA Augment Second Dose: This trial was a single-dose, single-arm, open-label trial. The only treatment arm was a percutaneous injection of NKA.
Arm/Group | NKA Augment Second Dose
Number analyzed (Participants) | 1
Age, Customized [Count of Participants; unit: Participants] — 59 years of age measured from birth.
  Participants
    59 years old | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Procedure and/or Product Related Serious Adverse Events (AE's) Through 12 Months Following the Final NKA Implantation
Description: Procedure and/or product related adverse events (AE's) through 12 months following the final NKA implantation, as measured by AE reporting.
Time Frame: 12 months following final implantation
Measure: Number; unit: Serious adverse events
Units Other Than Participants: Adverse events
Arm/Group | NKA Augment Second Dose
Number analyzed (Participants) | 1
Number analyzed (Adverse events) | 18
Serious adverse events | 2

2. Primary Outcome: Serial Estimation of Glomerular Filtration Rate (GFR) Through 6 Months Following the Final Cell Implantation, as Measured by Serial Serum Creatinine.
Description: The patient's serum creatinine was measured using a blood test at predetermined intervals and used to estimate the glomerular filtration rate as an indication of overall renal function.
Time Frame: 6 months following final cell implantation
Population: The single patient enrolled in the study was analyzed.
Measure: Number; unit: mL/min/1.73 m2
Groups:
- Neo-Kidney Augment: NKA was made from expanded autologous selected renal cells (SRC) obtained from the patient's kidney biopsy. To manufacture NKA, kidney biopsy tissue from each enrolled patient will be sent to RegenMedTX, LLC, where renal cells will be expanded and SRC selected. SRC will be formulated in a gelatin based hydrogel at a concentration of 100 x 106 cells/mL, packaged in a 10 mL syringe, and shipped to the clinical site for use.
Arm/Group | Neo-Kidney Augment
Number analyzed (Participants) | 1
mL/min/1.73 m2
  Baseline eGFR | 14
  Final eGFR | 11

3. Secondary Outcome: Renal-specific Laboratory Assessments Through 12 Months Following the Last NKA Implantation Under This Protocol.
Description: Renal-specific laboratory assessments through 12 months following the last NKA implantation under this protocol, whether first or second, as measured by renal specific biomarkers.
Time Frame: 12 months following last NKA implantation under this protocol
Population: Biomarkers were not analyzed for the one subject enrolled. There are no data for this outcome.
Arm/Group | Neo-Kidney Augment
Number analyzed (Participants) | 0

4. Other Pre Specified Outcome: Laboratory Assessments of Renal Function
Description: Laboratory assessments of renal function (including eGFR, serum creatinine, and proteinuria) to assess changes in the rate of progression of renal disease; and effect of method of implantation on these parameters.
Time Frame: 12 months following initial NKA implantation
Population: These data were not analyzed for the one patient enrolled.
Arm/Group | Neo-Kidney Augment
Number analyzed (Participants) | 0

5. Other Pre Specified Outcome: Quality of Life as Measured by Serial Kidney Disease Quality of Life Surveys
Description: Quality of life as measured by serial Kidney Disease Quality of Life survey obtained at baseline and at 1, 3, 6, 7, 9, 12, 15 and 18 months after a patient's first NKA implantation.
Time Frame: Through 18 months after first NKA implantation
Population: Quality of life data were not analyzed for the one patient enrolled.
Arm/Group | Neo-Kidney Augment
Number analyzed (Participants) | 0

6. Other Pre Specified Outcome: Evaluation of Renal Structure Over Time as Measured by Imaging Modalities.
Description: Evaluation of renal structure over time as measured by imaging modalities including MRI and Scintigraphy.
Time Frame: 12 months following initial NKA implantation
Population: The data for the lone subject were not formally analyzed.
Arm/Group | Neo-Kidney Augment
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 296 days.
Arm/Group | NKA Augment Second Dose
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 1/1
Other Adverse Events (participants affected / at risk) | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NKA Augment Second Dose (N=1)
Worsening hypertension (Cardiac disorders) | 1 (1) — The event of worsening hypertension was attributed to the subject's omission of his usual morning dose of anti-hypertensive medications prior to the procedure. Furthermore, it is likely that the subject's post-procedural pain contributed .
Surgical pain of the left kidney (Surgical and medical procedures) | 1 (1) — Post-procedural pain was worse than anticipated, due to technically difficulty, retroperitoneal scarring related to the previous laparoscopic NKA injection two years earlier, and a large cyst which made maneuvering the injection needles difficult.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NKA Augment Second Dose (N=1)
Worsening of hyperparathyroidism (Endocrine disorders) | 1 (1)
Worsening of chronic kidney disease (Renal and urinary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-28): https://cdn.clinicaltrials.gov/large-docs/63/NCT02525263/Prot_SAP_000.pdf